CLINICAL TRIAL: NCT05940467
Title: Acute Sleep Loss and Arterial Stiffness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Daniel Patterson, PhD, NRP, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY23030068
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Arterial Stiffness

STUDY DESIGN:
Intervention Model Description: This is a prospective study whereby participants undergo periods of sleep loss
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Loss (Experimental): Participants will undergo a night shift work like schedule and be monitored with non-invasive devices while at-home (at set intervals) and during an in-lab phase (hourly) during a 97 continuous-hour protocol. During the in-lab phase, which is approximately 48 continuous hours, participants will undergo a 24-hour period of sleep loss, followed by a brief opportunity for an in-lab sleep opportunity of 5 hours, followed by another period of 19 hours of sleep loss before returning home for at-home monitoring. Measures of interest include arterial stiffness as measured by pulse wave velocity (PWV) and changes in subjective ratings (e.g., fatigue and sleepiness). Other measures include cognitive performance, total sleep during the protocol, and sleep depth during an in-lab sleep opportunity.
  Interventions: Other: Sleep Loss

INTERVENTIONS:
Other: Sleep Loss — Participants will undergo periods of sleep loss in a laboratory setting and be monitored hourly for changes in indicators of arterial stiffness (i.e., pulse wave velocity).

SUMMARY:
The overarching goal of this study is to mimic a night shift work like schedule and characterize circadian variation in Pulse Wave Velocity (PWV), a measure of arterial stiffness, and determine the impact of acute loss of sleep like that experienced by shift workers on PWV.

DETAILED DESCRIPTION:
Night shift work is associated with increased risk of cardiovascular disease (CVD). Pulse wave velocity (PWV) is a commonly used non-invasive measure of arterial stiffness and is strongly associated with CVD. Previous research links sleep loss, like that experienced by shift workers, to elevated levels or abnormal levels of PWV. In addition, there is some research that shows circadian variation in PWV, which has implications for future studies and when PWV should be assessed. The overarching goal of this study is to characterize circadian variation in PWV and determine the impact of acute loss of sleep on PWV during a schedule like that experienced by night shift workers.

ELIGIBILITY:
Inclusion Criteria:

An individual may be eligible to participate if they meet the following criteria:

1. are between the ages of 20 and 29 years;
2. have not been diagnosed or told by a healthcare clinician that they have a medical condition that may impact their blood pressure or cardiovascular health/system;
3. can abstain from smoking tobacco or chewing tobacco products;
4. can abstain from caffeine and exercise for 4 days in a row;
5. are not prescribed medications or take over the counter medications that may impact blood pressure or heart rate (a team physician will review any reported medications identified during screening);
6. do not have a physical condition that may interfere with using the upper arm, upper thigh, or access to the neck area for purposes of performing non-invasive measures linked to this protocol; and
7. feel that they can avoid working and complete the 4 day protocol without interruption.

Exclusion Criteria:

An individual will be excluded if they report:

1. a medical condition or diagnosis that may impact their blood pressure or heart rate;
2. taking any standing medications or prescriptions, other than over the counter medications or contraceptives, that may impact their blood pressure or heart rate;
3. are unable to adhere to a strict 4 day protocol that involves abstaining from caffeine, alcohol, tobacco products (nicotine), and exercise;
4. have a physical condition that may limit use of the upper arm or upper thigh or area around the neck, which is necessary for performing multiple non-invasive measures associated with this protocol.
5. being pregnant.

Because participants may awaken during the in-lab sleep opportunity when staff use the Sphygmocor device, it is important that staff and the study team know if the participant has ever experienced the following:

A] Sleep Paralysis; B] Night Terrors; C] Have Obstructive Sleep Apnea which requires the use of a CPAP Device; D] Become angry towards others when abruptly woken up; E] Become physical towards others when abruptly woken up.

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Circadian changes in pulse wave velocity (PWV) | Over 48 hours during in-lab phase.
  Circadian (day/night) variation in arterial stiffness as measured by pulse wave velocity (PWV) during the in-lab phase of the protocol during periods of sleep loss. Average PWV (in meters per second m/s) measures calculated over daylight hours compared to the average PWV measures calculated over nighttime hours.
Changes in pulse wave velocity (PWV) in response to 24 hours of acute sleep loss | First 24 hours of the in-lab phase of the study protocol.
  Arterial stiffness as measured by pulse wave velocity (PWV) in meters per second during the in-lab phase of the study protocol. The in-lab measurement compared to the 24th hour measurement.
Changes in pulse wave velocity (PWV) in response to 48 hours of acute sleep loss | 48 hours of the in-lab phase of the study protocol.
  Arterial stiffness as measured by pulse wave velocity (PWV) in meters per second during the in-lab phase of the study protocol. The first in-lab measurement compared to the 48th hour measurement.

OTHER OUTCOMES:
Sleepiness first 24 hours of acute sleep loss | First 24 hours of the in-lab phase of the study protocol.
  Changes in subjectively rated sleepiness in response to sleep loss using a single-item question with response options ranging from 0= Not At All to 5= Very Much. The first in-lab measurement compared to the 24th hour measurement.
Sleepiness at 48 hours of acute sleep loss | 48 hours of the in-lab phase of the study protocol.
  Changes in subjectively rated sleepiness in response to sleep loss using a single-item question with response options ranging from 0= Not At All to 5= Very Much. The first in-lab measurement compared to the 48th hour measurement.
Fatigue first 24 hours of acute sleep loss | First 24 hours of the in-lab phase of the study protocol.
  Changes in subjectively rated fatigue in response to sleep loss using a single-item question with response options ranging from 0= Not At All to 5= Very Much. The first in-lab measurement compared to the 24th hour measurement.
Fatigue at 48 hours of acute sleep loss | 48 hours of the in-lab phase of the study protocol.
  Changes in subjectively rated fatigue in response to sleep loss using a single-item question with response options ranging from 0= Not At All to 5= Very Much. The first in-lab measurement compared to the 48th hour measurement.
Pulse wave analysis first 24 hours of acute sleep loss | First 24 hours of the in-lab phase of the study protocol.
  Non-invasive measure of central augmentation index (as a percentage) will be assessed at set intervals during the protocol. The first in-lab measurement compared to the 24th hour measurement.
Pulse wave analysis at 48 hours of acute sleep loss | 48 hours of the in-lab phase of the study protocol.
  Non-invasive measure of central augmentation index (as a percentage) will be assessed at set intervals during the protocol. The first in-lab measurement compared to the 48th hour measurement.
Cognitive performance first 24 hours of acute sleep loss | First 24 hours of the in-lab phase of the study protocol.
  Cognitive performance as measured by the Psychomotor Vigilance Test Brief (PVT-B) as measured by lapses (reaction time >355ms). The first in-lab measurement compared to the 24th hour measurement.
Cognitive performance at 48 hours of acute sleep loss | 48 hours of the in-lab phase of the study protocol.
  Cognitive performance as measured by the Psychomotor Vigilance Test Brief (PVT-B) as measured by lapses (reaction time >355ms). The first in-lab measurement compared to the 48th hour measurement.
Sleep depth | As measured during the in-lab 5-hour sleep opportunity.
  Sleep depth as measured by portable electroencephalogram (EEG) and reported as total minutes of deep sleep during the in-lab sleep opportunity.
Total sleep duration | Total sleep duration (in minutes) during the entire protocol (over 97 hours).
  Total sleep duration (in minutes) as measured by wrist-worn actigraphy over the entire 97 hour study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Patterson, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not have a defined plan to share data with outside investigators.